CLINICAL TRIAL: NCT04956705
Title: Vitamin D and Calcium Supplementation at Danish Nursing Homes - Effects on Vitamin D Status and Physical Functioning
Brief Title: Vitamin D and Calcium Supplementation at Danish Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Charlotte Mortensen, Principal Investigator, University College Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Alias: 200462
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Frailty; Physical Disability; Aging; Muscle Weakness
MeSH Terms: conditions — Frailty; Muscle Weakness | interventions — Vitamin D; Calcium

STUDY DESIGN:
Intervention Model Description: The project estimates the impact of The Model for Improvement on implementing the recommendation of vitamin D and calcium supplementation at nursing homes. Furthermore, the project evaluates which effect an improved implementation can have on vitamin D status and physical functioning in nursing home residents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Model for Improvement (Experimental): Together with the health care staff at the nursing homes, the project group will identify which strategies to implement in order to increase the number of residents receiving the recommended daily supplements of 20 µg of vitamin D and 800-1000 mg of calcium. The Model for Improvement will be the methodological framework for defining, implementing, and evaluating strategies.
  Interventions: Dietary Supplement: Vitamin D and calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D and calcium — Either as tablets, droplets or sprays. Preferably daily doses of 20 µg of vitamin D and 800-1000 mg of calcium as recommended.

SUMMARY:
Nursing home residents are in high risk of vitamin D deficiency, which negatively affects bone health. Vitamin D and calcium supplements have shown to increase bone density and reduce fracture risk and may affect daily physical functioning. Therefore, The Danish Health Authority recommends all nursing home residents a daily supplement of 20 µg vitamin D and 800-1000 mg calcium. However, adherence to the recommendation is low.

The present project hypothesizes that this low adherence results in a high number of residents with a deficient or insufficient vitamin D status, and that daily physical functioning can be improved or maintained by an improved adherence to the recommendation.

DETAILED DESCRIPTION:
Background: Residents in nursing homes belong to one of the high-risk groups when it comes to vitamin D deficiency, which is associated with increased risk of osteoporosis, muscle weakness and generally decreased physical functioning and frailty. Therefore, the Danish Health Authority recommends that all residents in nursing homes receive a daily supplement of 20 µg of vitamin D in addition to 800-1000 mg of calcium. Some systematic reviews and meta-analyses find that daily supplementation of 20 µg of vitamin D can improve physical functioning and muscle strength among older adults, whereas others do not find an effect. However, most studies are performed in non-institutionalized older adults.

An online survey conducted in May 2020 has revealed that the recommendation of giving residents in nursing homes a daily supplement of 20 µg vitamin D and 800-1000 mg calcium is not routine clinical practice in Denmark. The Danish Health Authority highlights The Model for Improvement as a tool to use when working with evidence-based practice within prevention and health promotion in the municipalities.

Objectives:

* To increase use of the recommended supplements with vitamin D and calcium among residents at nursing homes using The Model for Improvement as a methodological tool.
* To investigate the effect of improved vitamin D and calcium supplement use on vitamin D status and daily physical functioning among residents at nursing homes.

Hypotheses:

* Vitamin D status among residents at nursing homes are low and the majority can be defined as vitamin D insufficient.
* Vitamin D status and daily physical functioning of the residents are positively affected by an improved implementation of the recommendation.

Design and Methods: The project has a quasi-experimental design without control groups. It estimates the causal impact of The Model for Improvement on implementing the specific recommendation in a realistic setting at the nursing homes.

The study includes the following endpoints related to the older adults at the nursing homes evaluated before and after the intervention:

* Number of residents at the participating nursing homes taking supplementation of ≥20 µg of vitamin D and/or ≥800 mg of calcium ≥5 days/week.
* Number of residents at the participating nursing homes classified as having an insufficient and deficient vitamin D status (serum 25-hydroxyvitamin D (25(OH)D <50 nmol/L and <25 nmol/L, respectively)
* Mean daily physical functioning measured as muscle strength, 30-s chair-stand test, and a timed-up-and-go test.

ELIGIBILITY:
Inclusion Criteria:

* Being a resident at the participating nursing homes
* Understand and speak Danish in order to understand the study procedures
* Be able to give informed consent

Exclusion Criteria:

* Having kidney diseases
* Receiving medication which may induce adverse effects in combination with vitamin D and/or calcium supplements
* Being terminally ill
* Declared incompetent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of residents having vitamin D and calcium supplements daily | 6 months
  Assessed as those having ≥ 20 µg vitamin D and/or ≥ 800 mg calcium ≥ 5 days /week

SECONDARY OUTCOMES:
Vitamin D status | 6 months
  Assessed as 25-hydroxyvitamin D
Handgrip strength | 6 months
  Assessed with a digital handgrip dynamometer
Physical functioning | 6 months
  Assessed with timed-up-and-go test and 30-s chair-stand test

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Mortensen, PhD, Principal Investigator — University College Copenhagen
Locations (2):
- Denmark (2):
  - Frederiksgadecenteret, Haslev
  - Plejecentret Solbakken, Ringsted

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortensen C, Beck AM, Tetens I, Jeppesen C, Jorgensen SF, Nielsen LK, Kristensen M. Vitamin D Status and Physical Functioning in Nursing Home Residents after Improved Adherence to the Vitamin D and Calcium Recommendation-A Quasiexperimental Study. J Nutr Metab. 2024 Oct 5;2024:2405429. doi: 10.1155/2024/2405429. eCollection 2024. PMID 39398329